CLINICAL TRIAL: NCT01564771
Title: Serotype Distribution of Chest X-ray Confirmed Pneumococcal Community Acquired Pneumonia in the Adult Population in Greece, Over 1 Year.
Acronym: B1851065
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851065
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Pneumococcal Disease
Keywords: Pneumococcal serotypes; Community Acquired Pneumonia (CAP)
MeSH Terms: conditions — Pneumococcal Infections; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group one: Adults ≥18 years of age with chest X-ray confirmed CAP
  Interventions: Other: Non Intervention

INTERVENTIONS:
Other: Non Intervention — This Is A Non Interventional Study

SUMMARY:
Serotype distribution and estimation of antimicrobial resistance in S. pneumoniae isolates and anticipated PCV7 and PCV13 coverage is difficult in Greece, because invasive isolates collected each year are limited and depict a certain proportion of patients who have easy access to tertiary care or have underlying medical reasons which necessitate inpatient care. It is also probable that the real burden of pneumococcal disease is not well estimated especially among adults. New additions in the laboratory setting such as the pneumococcal urine antigen assay (Binax NOW®) and the Urinary Antigen Diagnostic Assay (Luminex) for the detection of 13 serotype specific polysaccharides in human urine developed by Pfizer might be helpful in identifying more pneumococcal infections compared to the previous years. This NIS is based on the unmet scientific need to describe the serotype distribution and the resistance profile of isolates from X-Ray confirmed CAP in the present circumstances.

DETAILED DESCRIPTION:
For each surveillance period lasting for 12 months all adults presenting in the selected clinics with symptoms and signs suggestive of pneumonia (candidate cases) will be asked to participate in the study

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in the study and agreed to sign an ICD.
* Patients had to be ≥18 years of age (adults)
* Patients had to present or had been referred to a participating healthcare facility with suspected pneumonia based on the physician's assessment (including but not limited to specific signs and symptoms described in Section 9.3 of the protocol)
* Patients must have had a posteroanterior or anteroposterior chest X-ray showing an infiltrate (if previous films were not available) or a new infiltrate (if recent film was available)
* Patients had to be tested positive for the Binax NOW® assay (required post Protocol Amendment 2)

Exclusion Criteria:

* Patients who did not sign an ICD.
* Any patient who developed signs and symptoms of pneumonia after being hospitalized for ≥48 hours
* Any patient who was transferred to a study healthcare facility after already being hospitalized for ≥48 hours at another healthcare facility
* Patients who did not have a chest X-ray performed
* Patients who did not have the Binax NOW® assay performed
* Patients with negative results for the Binax NOW® assay (required post Protocol Amendment 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults ≥18 years of age with chest X-ray confirmed CAP
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The frequency of serotypes 4,6B,9V,14,18C,19F,23F,1,3,5,6A,7F and 19A from chest X-ray confirmed pCAP patients (post amendment2 with positive Binax NOW® only) who presented in the emergency departments of 15 hospitals in Greece during 1 | One year
calendar year. | One year

SECONDARY OUTCOMES:
Susceptibility, resistance or partial resistance Streptococcus pneumoniae clinical isolates obtained from study adult CAP patients. | One year
The frequency of the 4, 6B, 9V, 14, 18C, 19F, 23F, 1, 3, 5, 6A, 7F, 19A serotypes (based on Luminex assay) of study patients immunized and not immunized with PPV. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (21):
- Greece (21):
  - General Hospital of Athens "Evangelismos" / Pneumonology Department, Athens, Attica
  - University Hospital of Alexandroupolis, Alexandroupoli, Evros
  - General University Hospital of Alexandroupoli, Alexandroupoli
  - General Chest Diseases Hospital "Sotiria"/ 7th Department of Pulmonary Medicine, Athens
  - General Hospital of Athens "Sotiria"/ 12Th Pneumonology Clinic, Athens
  - General Hospital of Athens "Sotiria"/ 1St Pneumonology Clinic, Athens
  - General Hospital of Athens "Sotiria"/ 2Nd Pneumonology Clinic, Athens
  - General Hospital of Athens "Sotiria"/ 5Th Pneumonology Clinic, Athens
  - General Hospital of Athens "Sotiria"/ 6Th Pneumonology Clinic, Athens
  - General Hospital of Athens "Sotiria"/ 8Th Pneumonology Clinic, Athens
  - Diagnostic Therapeutic Center of Athens Ygeia, Athens
  - General Hospital Athens "Sismanoglio"/ 1St Pneumonology Clinic, Athens
  - General Hospital of Athens "Sismanoglio" / 3Rd Pneumonology Department, Athens
  - General Hospital of Athens "Sismanoglio"/ 2Nd Pneumonology Clinic, Athens
  - General Hospital Mellision "Amalia Fleming"/ Pneumonology Clinic, Athens
  - General Hospital Mellision "Amalia Fleming"/2nd Internal Medicine Department, Athens
  - Sotiria Hospital, Intensive Care Unit, Athens
  - General University Hospital "Attikgeneral University Hospital "Attikon"/ 4Th University Internal Med, Athnens
  - General Hospital of Kavala/ A Pneumonological Clinic, Kavala
  - General Hospital of Kavala/ b Pneumonological & Tubeculosis Department, Kavala
  - University General Hospial of Larissa, Pneumonology Department, Larissa

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851065&StudyName=Serotype%20Distribution%20of%20Chest%20X-ray%20Confirmed%20Pneumococcal%20Community%20Acquired%20Pneumonia%20%20in%20the%20Adult%20Population%20in%20Greece%2C%20Over%201%20Ye